CLINICAL TRIAL: NCT04102241
Title: A Phase Ⅱ Efficacy and Safety Study of Hemay005 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy and Safety Study of Hemay005 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM005PS2S01
Record Dates: First submitted 2019-03-20; First posted 2019-09-25 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Psoriasis
Keywords: psoriasis; PDE4
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Patients with chronic plaque psoriasis will be treated BID for 16 weeks with placebo in first phase. Then will be treated BID for 36-week extension followed with 30mg of Hemay005.
  Interventions: Drug: Placebos
- 15mg Hemay005 (Experimental): Patients with chronic plaque psoriasis will be treated BID for 16 weeks with 15mg Hemay005 in first phase. Then will be treated BID for 36-week extension followed with 15mg of Hemay005.
  Interventions: Drug: 15mg Hemay005; Drug: Placebos
- 30mg Hemay005 (Experimental): Patients with chronic plaque psoriasis will be treated BID for 16 weeks with 30mg Hemay005 in first phase. Then will be treated BID for 36-week extension followed with 30mg of Hemay005.
  Interventions: Drug: 15mg Hemay005; Drug: Placebos
- 60mg Hemay005 (Experimental): Patients with chronic plaque psoriasis will be treated BID for 16 weeks with 60mg Hemay005 in first phase. Then will be treated BID for 36-week extension followed with 60mg of Hemay005.
  Interventions: Drug: 15mg Hemay005

INTERVENTIONS:
Drug: 15mg Hemay005 — Hemay005 is a small molecule PDE4 inhibitor.
  Other Names: No other intervention name.
  Arms: 15mg Hemay005; 30mg Hemay005; 60mg Hemay005
Drug: Placebos — Placebos are the same as drugs, but contain no Hemay005.
  Other Names: No other intervention name.
  Arms: 15mg Hemay005; 30mg Hemay005; Placebo

SUMMARY:
Hemay005 is a novel phosphodiesterase type 4(PDE4) inhibitor being developed for the treatment of psoriasis.After single asending dose and mutiple asending dose in health subjects. And the patients with moderate to severe plaque psoriasis will be randomized into 4 cohorts(15mg, 30mg, 60mg and placebo) approximately 216 subjects will be enrolled (52 for each cohort ). This study includes an 16-week treatment Period, then a 36-week Treatment Period without placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age and less than or equal to 75;
* Diagnosed with plaque psoriasis more than 6 months;
* Screening and baseline PSAI ≥12, sPGA≥3（Moderate to Severe）,affected body surface area BSA≥10%;
* Investigator determined suitable for systemic treatment of psoriasis;
* All subjects must agree and commit to the use of a reliable contraceptive regimen. Women of childbearing potential must undergo monthly pregnancy testing during the study and agree to use two of the following methods of contraception throughout the study and for 90 days after the last dose of study drug. Reliable contraceptive regimen: vasectomy, abstinence, the use of condoms, intrauterine contraceptives (IUD), (Oral administration, patch, ring, injection, implantation) Barrier methods (diaphragm with spermicide, condom with spermicide);
* Ability to understand and be willing to sign a written informed consent before study entry.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type; (i.e., erythrodermic and guttate psoriasis, palmar, plantar or nail disease) at screening, Investigator diagnosed with drug-induced psoriasis (i.e., from beta-blockers, calcium channel inhibitors or lithium) prior to randomization;
* A history of chronic infection (i.e., tuberculosis);
* A condition of any skin disease(i.e., dermatitis) ;
* History of systemic autoimmune inflammatory disease that effect drug evaluation;
* Patients with an active infection who are assessed by the investigator as at increased risk;
* TB infection, high risk of acquiring TB infection, latent TB infection (LTBI), or current or history of NTMB infection;
* Subjects who used any of the following treatments : 2 weeks before randomize (including but not limited to local use of Glucocorticoids, topical retinoic acid preparations, vitamin D derivatives, tacrolimus, pimeklimus, dianthranol, etc) Except for the following situations: In the face, armpit and groin psoriasis skin lesions using weak or inefficient local use of glucocorticoid (efficacy grade 6-7) or scalp psoriasis skin lesions with coal tar shampoo, salicylic acid topical preparations, selenium disulfide, the use of non-pharmaceutical emollients (such as silicone cream, vitamin E cream, etc.) ; 4 weeks before randomize , Non-biological drug systemic therapy (including but not limited to systemic glucocorticoid, leflunomide, cyclophosphamide, methotrexate, cyclosporine, retinoic acid, traditional Chinese medicine decoction, proprietary Chinese medicine for the treatment of psoriasis, etc.), 2 weeks before randomize with UVB treatment, 4 weeks before randomize with psoralen and long wave ultraviolet (PUVA) therapy, 12 weeks before randomize with biological agents such as adamuzumab, enasip or infliximab, 24 weeks before randomize with alefacept, Briakinumab, Ustekinumab, Secukinumab; Subjects with psoriasis worsen or rebound 4 weeks before screening;
* Subjects who congenital or acquired immunodeficiency;
* Subjects couldn't limit their uv exposure during the study period (e.g. sunbathing and/or tanning devices);
* History of apremilast ;
* Subjects with conditions that may affect oral drug absorption, such as subtotal gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of weight-loss surgery, such as gastric bypass surgery, do not include surgery that simply separates the stomach into separate Chambers, such as gastric banding surgery;
* sCr≥1.5 upper limit of normal (ULN); AST≥2ULN; ALT≥2 ULN
* WBC<3.0×109/L or WBC>14×109/L,PLT<100×109/L, Hb<85 g/L;
* Subjects with a malignant tumor, or any history of malignancy within 5 years (except skin squamous cell carcinoma in situ, basal cell carcinoma or cervical carcinoma in situ that has been treated and has no evidence of recurrence in the past 12 weeks);
* Subjects with positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening;
* Has a history of alcohol or drug abuse or dependence, or a history of mental illness;
* Has committed suicide (Includes active attempts, discontinued attempts or attempted attempts) or suicidal thoughts within the past 6 months;
* Pregnant or lactating women or planning pregnancy during the study period;
* Know allergic to active ingredient or excipient of the investigational product;
* 4 weeks before randomize, participated in a clinical trial and use of the study drug;
* Accompanied by severe, progressive, or uncontrolled disease or in the investigator's opinion unsuitable to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have 75% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI75). | week16
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) at week 16.

SECONDARY OUTCOMES:
Severity of Adverse Events and Serious Adverse Events. | week2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56.
  Severity of all Adverse Events (AEs) and Serious Adverse Events (SAEs) that occur during the whole trial including the observational period (AEs and SAEs include but not limited to comorbidities, such as hypertension, diabetes, and cardiovascular diseases).
Cmax of Hemay005. | week8
  Maximum observed serum concentration.
Proportion of subjects achieving an overall sPGA score of clear (0) or almost clear (1) with at least a 2-point reduction from baseline. | week2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56.
  The static Physician's Global Assessment (sPGA) rated the investigator's overall clinical assessment of a participants plaque thickness, erythema, and scaling on a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (majority of plaques have severe thickness, erythema, and scale). To assign a sPGA score, the investigator examined all psoriatic lesions and assigned a severity score ranging from 0 to 5 for thickness, erythema, and scaling. Scores for thickness, erythema, and scaling are summed and the mean of these 3 scores equals the overall sPGA score. Decreases in sPGA correspond to clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, Dr, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China